CLINICAL TRIAL: NCT07149389
Title: A Clinical and Epidemiological Study of Children With Acute Respiratory Distress Presenting to the Emergency Unit at Assiut University Children Hospital, Egypt
Brief Title: Assessment of Acute Respiratory Distress in Children Presenting to the Emergency Department: Clinical, Epidemiological, and Etiological Insights
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma Ayman, resident at the pediatrics department, Assiut University
Other Study IDs: Children with ARD
Record Dates: First submitted 2025-08-28; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: acute respiratory distress; ARD
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- acute respiratory distress patients: Children aged between 1 month and 18 years presenting with acute respiratory distress at the emergency department of Assiut University Children Hospital are studied

SUMMARY:
This study investigates the clinical and epidemiological characteristics of children with acute respiratory distress presenting to the emergency unit at Assiut University Children Hospital. It aims to determine the prevalence, causes, and risk factors to improve understanding and management of this critical pediatric condition.

DETAILED DESCRIPTION:
This descriptive cross-sectional study will be conducted over six months in the pediatrics emergency department of Assiut University Hospital, Egypt. It enrolls children aged 1 month to 18 years presenting with acute respiratory distress (ARD). The study collects detailed demographic, clinical, environmental, nutritional, and developmental data using a structured, pre-tested case record form. It includes comprehensive patient history, physical examination, laboratory and radiological investigations to identify underlying causes, clinical features, and risk factors for ARD. Data will be analyzed statistically using SPSS software to characterize the epidemiology and clinical spectrum, inclusion of factors like exposure to passive smoking, socioeconomic status, and detailed symptomatology, aiming to contribute to better diagnosis, treatment, and prevention strategies in this resource-limited setting

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 month to 18 years
* children presenting to the emergency department with acute respiratory distress.

Exclusion Criteria:

* Patients older than 18 years or younger than 1 month.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population consists of pediatric patients from urban and rural areas of Upper Egypt who seek emergency care for acute respiratory distress. The cohort reflects diverse socioeconomic backgrounds, maternal education levels, and environmental exposures such as household air quality and passive smoking. The children present with various severities of respiratory distress caused by multiple etiologies including pulmonary, cardiac, infectious, metabolic, and neurological factors. Nutritional assessments and developmental milestones are documented as potential modifiers of disease presentation and outcomes. Comprehensive laboratory tests and imaging help confirm diagnoses and severity, with particular attention to those at higher risk of complications. As such, this population offers a representative sample of pediatric ARD patients in a regional tertiary care center.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2026-08-30 (Estimated); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute respiratory distress among children | Baseline
  Measurement of how frequently ARD occurs in children presenting at the emergency department

REFERENCES:
- [Background] Kango SC, Yanza MCAS, Komba JEK, Mand&#233 M, -Njapou, Gody JC, et al. Epidemiological, Clinical and Therapeutic Aspects of Acute Respiratory Distress in Children in Medical Emergencies at the Bangui Pediatric University Hospital. Open J Pediatr 2025;15:111-8. https://doi.org/10.4236/OJPED.2025.151011.